CLINICAL TRIAL: NCT01071863
Title: Association of Fear of Falling and Physical Activity in Rheumatoid Arthritis Comparison Before and After Biological Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Dr David Walker, Newcastle upon Tyne hospitals NHS Foundation Trust
Other Study IDs: RA-FOF-ACT-2010
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2010-02-22 (Estimated); Status verified 2010-02

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rheumatoid Arthritis (RA) Patient Group: Patients with RA who have been refered for biological drug treatment
- Control Group: 20 people of same age and sex as the RA patient cohort

SUMMARY:
Primary Objective:

To identify the prevalence and severity of the fear of falling in a rheumatoid population

Secondary Objectives:

To explore the effect the treatment with biological agents has on fear of falling and physical activity in a rheumatoid population

DETAILED DESCRIPTION:
The study will be an open, observational study to determine the prevalence of fear of falling in a rheumatoid population with severe disease being considered for biological therapy; this will be compared with physical activity levels at baseline and the change in these level pre and post treatment with biologic therapy. An age and sex matched control group will also be studied to allow inference to be drawn from the self reported 'fear of falling' and the objective activity levels of the RA population.

The study will consist of two visits: screening/baseline, and a 12 week follow up visit. It will be an observational study of the effects of the planned treatment regime via the NHS pathway. The subjects who are eligible to enter in the study will receive his/her normal treatment prescribed and be at the referral phase for biological treatment. The control group will continue on any existing treatments but will not have any reported physical limitations.

At the screening/baseline visit the self completion outcome questionnaires will be given to both the patient group and the control group. A disease activity score (aggregate score of RA symptoms - DAS) for the RA population will be calculated by a nurse specialist at the time of referral for the biological agent and again at 12 weeks post treatment, these parameters will not be repeated by the research team but the DAS score will be collected used in the final analysis. In addition, the Numact ambulatory activity recorder - used to assess spontaneous ambulatory activity - will be fitted for a 24hour period. This screening / baseline visit will occur before, but as near as possible to the 1st treatment day of the prescribed biological agent.

Occasionally the recording device may fail due to extraneous factors; in this instance a second recording may be required.

The control group will complete their study participation immediately after the screening / baseline visit.

The participant will then follow the care pathway of their treating physician with no interception by the study team. The 2nd and final study visit will be scheduled for 12 weeks post treatment with the biologic agent.

At 12 weeks a repeat assessment of the screening procedures will be made. Beyond which there will be no further study contact with the patients unless they request further discussion about the study findings. If they request this an appointment will be made at the time of the final study report/write up.

Physical examination could be carried out at any time during the study period if considered appropriate by the physician, however, this is not a predicted study procedure..

Details of any changes in medication and adverse events will be reported by subjects at the final visit, week 12.

ELIGIBILITY:
Inclusion criteria RA population:

1. Male and female subjects
2. Subjects with a clinical diagnosis of Rheumatoid Arthritis who have been referred for a biologic treatment
3. Subjects who are willing to complete the questionnaires and wear the Numact activity monitor
4. Written informed consent

Inclusion criteria Control group:

1. Male and female subjects
2. Age and sex matched to RA population (any appropriate sibling will be invited possibly siblings)
3. Subjects who are willing to complete the questionnaires and wear the Numact activity monitor
4. Written informed consent

Exclusion criteria RA Population:

1. Diagnosis or evidence of any other physically limiting condition
2. Subjects who have received an intramuscular steroid injection within 2 months of study entry or in whom such treatment is planned within the study period
3. Subjects scheduled for elective surgery of the disease site or any other elective major surgery which would fall within the study period
4. Subjects who currently abuse alcohol or drugs, or have a recent history of alcohol or drug abuse, or who in the Investigator's opinion, have previously demonstrated drug-seeking behavior
5. Subjects who are currently participating in another clinical research study involving a new chemical entity or who have participated in a clinical study within the previous 30 days
6. Subjects who the Investigator believes are unsuitable for the study

Exclusion criteria Control Group:

1. Diagnosis or evidence of any physically limiting condition
2. Subjects who currently abuse alcohol or drugs, or have a recent history of alcohol or drug abuse, or who in the Investigator's opinion, have previously demonstrated drug-seeking behavior
3. Subjects who the Investigator believes are unsuitable for the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20 patients with Rheumatoid arthritis refered for biological treatment 20 control subjects matched for age and sex
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-10 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
To identify the prevalence and severity of the fear of falling in a rheumatoid population

SECONDARY OUTCOMES:
To explore the effect the treatment with biological agents has on fear of falling and physical activity in a rheumatoid population

CONTACTS AND LOCATIONS:
Overall Officials: David J Walker, MD, Principal Investigator — Newcastle upon Tyne NHS Foundation Trust
Locations (1):
- Newcastle upon Tyne NHS F Trust, Newcastle, UK, United Kingdom